CLINICAL TRIAL: NCT02550860
Title: Influence of Fish Oil Based Intravenous Fat Emulsions on the Epidermal Barrier Function
Acronym: Tewlip
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: problem of enrollment
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-786
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Intestinal Diseases
Keywords: intravenous fat emulsions; parenteral nutrition; skin barrier function; essential fatty acids; transepidermal water loss
MeSH Terms: conditions — Intestinal Diseases; Hyperphagia | interventions — Soybean Oil; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- soybean oil (SO)-based IVFE (Medialipide) (Active Comparator)
  Interventions: Drug: soybean oil (SO)-based IVFE (Medialipide)
- fish oil (FO)-containing IVFE (Lipidem) (Active Comparator): fish oil (FO)-containing IVFE (Lipidem)
  Interventions: Drug: fish oil (FO)-containing IVFE (Lipidem)

INTERVENTIONS:
Drug: soybean oil (SO)-based IVFE (Medialipide) — The soybean oil (SO)-based IVFE will be allocated for a 3-month period, allowing sufficient timeframe for epidermal complete renewal.
  Arms: soybean oil (SO)-based IVFE (Medialipide)
Drug: fish oil (FO)-containing IVFE (Lipidem) — The fish oil (FO)-containing IVFE will be allocated for a 3-month period, allowing sufficient timeframe for epidermal complete renewal.
  Arms: fish oil (FO)-containing IVFE (Lipidem)

SUMMARY:
The epidermal barrier efficacy is determined by the physicochemical properties of the epidermal lipid matrix, among which ω-6 essential fatty acids (EFAs) play a key role. Inversely, the ω-3 EFAs are not found in the epidermis. For patients receiving lipid-containing parenteral nutrition (LCPN), the improvement of the epidermal barrier through the infusion of most appropriate intravenous fat emulsions (IVFE) could have many applications in clinical nutrition, mainly limiting water loss in patients receiving long-term LCPN and help in electrolyte and water balance.

The objective of this interventional clinical trial is to evaluate the epidermal barrier function in patients receiving long-term LCPN comparing two compositions of IVFE: (i) soybean oil (SO)-based IVFE (Medialipide) or (ii) fish oil (FO)-containing IVFE (Lipidem). Epidermal barrier function will be assessed through the transepidermal water loss (TEWL) measurement on the skin surface, a validated marker of the epidermal barrier efficacy. The two IVFE (SO-based or FO-containing) will be compared using a randomized double blind crossover design, using patients as their own control. Each IVFE will be allocated for a 3-month period, allowing sufficient timeframe for epidermal complete renewal. Patient's epidermal and red blood cell EFA profile will be determinate in order to facilitate result interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sever chronic intestinal disease requiring long term parenteral nutrition
* Receiving home lipid containing parenteral nutrition (LCPN), regardless of currently infused intravenous fat emulsion
* With a stable dose of LCPN for at least 1 month at recruitment time
* Administered at least 4 days a week through central venous access, with at least 150 mL of lipid per parenteral nutrition bag with lipid.
* Age >18
* Being available for 2 medical consultations in a 6 month period
* Who gave its written informed consent to participate to the study and without legal protection
* Social security coverage

Exclusion Criteria:

* Lesser expected parenteral nutrition length than duration for the entire trial
* Dermatological criteria : History of skin disease (atopic dermatitis, psoriasis) or evolving skin disease, broken or inflamed skin on the TEWL measurement site, Use of topical creams on the TEWL measurement site, Skin or systemic allergy (asthma)
* Contraindication to one of the selected intravenous fat emulsion: Severe dyslipidemia; Uncontrolled diabetes; Sepsis; Severe hepatic impairment; Major blood clotting disorders; Egg protein, soybean, peanut or fish hyper sensibility; Serum creatinine clearance < 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the transepidermal water loss (TEWL). | at Day 0 (at recruitment time)
  Measurement will be performed in a horizontal plane on the dominant volar forearm, which is the reference site for TEWL measurement because of its low content of sebaceous glands and pilosity. The TEWL will be measured using the latest generation of closed chamber system, combined to a vapor water condenser (Aquaflux 200®), which offers the advantage of a reduced TEWL value sensitivity to ambient humidity and temperature during measurement.
Measurement of the transepidermal water loss (TEWL). | at Day 90
  Measurement will be performed in a horizontal plane on the dominant volar forearm, which is the reference site for TEWL measurement because of its low content of sebaceous glands and pilosity. The TEWL will be measured using the latest generation of closed chamber system, combined to a vapor water condenser (Aquaflux 200®), which offers the advantage of a reduced TEWL value sensitivity to ambient humidity and temperature during measurement.
Measurement of the transepidermal water loss (TEWL). | at Day 180
  Measurement will be performed in a horizontal plane on the dominant volar forearm, which is the reference site for TEWL measurement because of its low content of sebaceous glands and pilosity. The TEWL will be measured using the latest generation of closed chamber system, combined to a vapor water condenser (Aquaflux 200®), which offers the advantage of a reduced TEWL value sensitivity to ambient humidity and temperature during measurement.

SECONDARY OUTCOMES:
Determination of erythrocyte fatty acids ω-6 | at Day 0
  Essential fatty acid red blood cell monitoring more properly reflect the global membrane fatty acid composition of the body. Monitoring will be achieved at biochemistry laboratory of recruiting centers on a blood sample.
Determination of erythrocyte fatty acids ω-3 | at Day 0
  Essential fatty acid red blood cell monitoring more properly reflect the global membrane fatty acid composition of the body. Monitoring will be achieved at biochemistry laboratory of recruiting centers on a blood sample.
Determination of erythrocyte fatty acids ω-6 | at Day 90
  Essential fatty acid red blood cell monitoring more properly reflect the global membrane fatty acid composition of the body. Monitoring will be achieved at biochemistry laboratory of recruiting centers on a blood sample.
Determination of erythrocyte fatty acids ω-3 | at Day 90
  Essential fatty acid red blood cell monitoring more properly reflect the global membrane fatty acid composition of the body. Monitoring will be achieved at biochemistry laboratory of recruiting centers on a blood sample.
Determination of erythrocyte fatty acids ω-6 | at Day 180
  Essential fatty acid red blood cell monitoring more properly reflect the global membrane fatty acid composition of the body. Monitoring will be achieved at biochemistry laboratory of recruiting centers on a blood sample.
Determination of erythrocyte fatty acids ω-3 | at Day 180
  Essential fatty acid red blood cell monitoring more properly reflect the global membrane fatty acid composition of the body. Monitoring will be achieved at biochemistry laboratory of recruiting centers on a blood sample.
Determination of Stratum corneum (SC) ω-3 | at Day 0
  Stratum corneum lipids will be collected using the minimally invasive and painless "Tape Stripping" method, which consists of applying a scotch on the skin. Quantitative and qualitative composition of the SC lipid matrix will be determined using high-performance thin-layer chromatography.
Determination of Stratum corneum (SC) ω-6 | at Day 0
  Stratum corneum lipids will be collected using the minimally invasive and painless "Tape Stripping" method, which consists of applying a scotch on the skin. Quantitative and qualitative composition of the SC lipid matrix will be determined using high-performance thin-layer chromatography.
Determination of Stratum corneum (SC) ω-3 | at Day 90
  Stratum corneum lipids will be collected using the minimally invasive and painless "Tape Stripping" method, which consists of applying a scotch on the skin. Quantitative and qualitative composition of the SC lipid matrix will be determined using high-performance thin-layer chromatography.
Determination of Stratum corneum (SC) ω-6 | at Day 90
  Stratum corneum lipids will be collected using the minimally invasive and painless "Tape Stripping" method, which consists of applying a scotch on the skin. Quantitative and qualitative composition of the SC lipid matrix will be determined using high-performance thin-layer chromatography.
Determination of Stratum corneum (SC) ω-3 | at Day 180
  Stratum corneum lipids will be collected using the minimally invasive and painless "Tape Stripping" method, which consists of applying a scotch on the skin. Quantitative and qualitative composition of the SC lipid matrix will be determined using high-performance thin-layer chromatography.
Determination of Stratum corneum (SC) ω-6 | at Day 180
  Stratum corneum lipids will be collected using the minimally invasive and painless "Tape Stripping" method, which consists of applying a scotch on the skin. Quantitative and qualitative composition of the SC lipid matrix will be determined using high-performance thin-layer chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Barnoud, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite